CLINICAL TRIAL: NCT02298049
Title: Satiation Attenuates BOLD Activity in Brain Regions Involved in Reward and Increases Activity in an Inhibitory Control Area: an fMRI Study in Healthy Volunteers.
Brief Title: An fMRI Study of Satiation in Healthy Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UBirmingham
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Appetite
Keywords: fMRI; reward; satiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scanning (Other): Repeated measures:
  Satiation scan + Pre-meal scan
  All participants undertook both scans
  Interventions: Other: Satiated / Pre-meal; Device: MRI

INTERVENTIONS:
Other: Satiated / Pre-meal — All participants were scanned before and after not being fed (pre-meal), and before and after being given a satiating lunch (satiated).
Device: MRI

SUMMARY:
To our knowledge no study has assessed the effects of a meal on neural responses to food cues and compared this with a condition simulating natural inter-meal hunger levels. This is important, as the existing literature often compares the effect of fasting to satiation, which may not reflect typical appetite processes. Thus, the purpose of this research was to examine the effect of a satiating lunch compared to a normal pre-meal state on blood oxygen level dependent (BOLD) activity in the human brain, as measured using functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
We hypothesized that satiation would be associated with decreased brain activity across brain regions involved in both appetite and reward such as ventromedial prefrontal cortex, orbitofrontal cortex, ventral striatum, hypothalamus, insula, amygdala and hippocampus. 16 healthy participants (8 males) were scanned on two separate test days, before and after eating a meal to satiation, or after not eating for 4 hours (satiated vs. pre-meal). fMRI BOLD signals to the sight and/or taste of the stimuli were recorded. Participants were given questionnaires to complete about their mood state and appetite before and after all scans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Sufficiently fluent in English to understand the task and the instructions

Exclusion Criteria:

* Currently taking medication
* Past or current depression/dieting,
* Smokers
* Food allergies
* Diabetes
* Pregnancy
* BMI score outside the normal range
* Any contraindications to fMRI scanning (e.g. pacemakers, mechanical heart valve, hip replacement, metal implants)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Activation differences between satiated and pre-meal scan fMRI BOLD signal | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Thomas, MRes, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Thomas JM, Higgs S, Dourish CT, Hansen PC, Harmer CJ, McCabe C. Satiation attenuates BOLD activity in brain regions involved in reward and increases activity in dorsolateral prefrontal cortex: an fMRI study in healthy volunteers. Am J Clin Nutr. 2015 Apr;101(4):697-704. doi: 10.3945/ajcn.114.097543. Epub 2015 Jan 21. PMID 25833968